CLINICAL TRIAL: NCT00251680
Title: A Placebo-Controlled, Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 100 mg in Subjects With Type 2 Diabetes Currently Treated With Lipid-Lowering Therapy
Brief Title: Efficacy of Lapaquistat Acetate in Subjects Currently Treated With Lipid-Lowering Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475/EC304; 2005-002316-24 (EudraCT Number); U1111-1122-8281 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Atorvastatin; Simvastatin; Rosuvastatin Calcium; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 50 mg QD (Experimental): (and stable lipid-lowering therapy)
  Interventions: Drug: Lapaquistat acetate and lipid-lowering therapy
- Stable Lipid-lowering therapy (Active Comparator)
  Interventions: Drug: Lipid-lowering therapy

INTERVENTIONS:
Drug: Lapaquistat acetate and lipid-lowering therapy — Lapaquistat acetate 50 mg, tablets, orally, once daily and stable lipid-lowering therapy for up to 24 weeks.
  Other Names: TAK-475; Lipitor; Zocor; Crestor; Tricor
  Arms: Lapaquistat Acetate 50 mg QD
Drug: Lipid-lowering therapy — Lapaquistat acetate placebo-matching tablets, tablets, orally, once daily and stable lipid-lowering therapy for up to 24 weeks.
  Other Names: Lipitor; Zocor; Crestor; Tricor
  Arms: Stable Lipid-lowering therapy

SUMMARY:
The purpose of the study is to determine the efficacy of lapaquistat acetate, once daily (QD), taken with established lipid-lowering therapy in subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus is a recognized cause of secondary dyslipidemia, and is also independently considered to be a major cardiovascular risk factor requiring aggressive lipid-lowering treatment. Type 2 diabetes accounts for 85% to 90% of diabetes worldwide. It affects about 2% of the Caucasian population in most Westernized countries, and the prevalence rises with age to 10% in those over 70 years of age. Five percent or more of young- and middle-aged adults in some Asian or Afro-Caribbean groups in the United Kingdom have this condition. Approximately 12 million Americans have type 2 diabetes, and an estimated 20 million more have some degree of glucose intolerance. The greatest cause of mortality in type 2 diabetes is atherosclerotic vascular disease and its sequelae between 75% and 80% of adult subjects with diabetes die of macrovascular complications.

Lapaquistat acetate is a squalene synthase inhibitor currently under development at Takeda for the treatment of dyslipidemia. This study will evaluate the efficacy and safety of lapaquistat acetate co-administered with an established lipid-lowering therapy including atorvastatin, simvastatin, rosuvastatin, or fenofibrate in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception from screening throughout the duration of the study and for 30 days following the last dose.
* Has a documented history of dyslipidemia with or without cardiovascular risk factors but without type 1 or 2 diabetes.
* Is on a stable antidiabetic regimen, which may have included oral antidiabetic medication and/or insulin, for at least 3 months prior to Screening.
* Prior to Randomization, the participant has a mean low density lipoprotein cholesterol level greater than or equal to 100 mg/dL and less than or equal to 190 mg/dL for 2 consecutive samples.
* Prior to Randomization, the subject has mean triglyceride level greater than or equal to 400 mg/dL for 2 consecutive samples.
* Is willing and able to comply with the recommended, standardized diet.

Exclusion Criteria:

* Has annine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, identified during screening.
* Has a serum creatinine greater than 133 mmol/L, identified during screening.
* Has a creatine kinase greater than 3 times the upper limit of normal, identified during screening.
* Has active liver disease or jaundice.
* Has taken any bile acid sequestrants [eg, cholestyramine], and intestinal cholesterol uptake inhibitors [eg, ezetimibe]) from 30 days before Screening until study completion or any fibrates for 6 weeks before Visit 1.
* Has a previous history of cancer that has been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, unstable angina, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary angioplasty, coronary or peripheral arterial surgery, or multiple risk factors that confer a 10-year risk for cardiovascular heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody test, as determined by medical history.
* Has a positive human immunodeficiency virus status or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has received any investigational medication 30 days prior to screening, or is participating in an investigational study.
* Has received lapaquistat acetate in a previous clinical study or as a therapeutic agent.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension
* Has had inflammatory bowel disease or any other malabsorption syndrome, or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of high alcohol intake within the previous 2 years.
* Has type 1 or 2 diabetes mellitus.
* Subject had a history of photoallergic or phototoxic reaction during treatment with a fibrate or ketoprofen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma Low Density Lipoprotein cholesterol | Week 24 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Triglycerides | Week 24 or Final Visit
Change from Baseline in Total Cholesterol | Week 24 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 24 or Final Visit
Change from Baseline in apolipoprotein B | Week 24 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 1.81 mmol/L (70 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 24 or Final Visit
Best corrected visual acuity | Week 24 or Final Visit
Adverse Events | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Clinical Laboratory Tests | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Vital Signs | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
12-lead Electrocardiogram | Weeks 12 and 24 or Final Visit
Physical Examination | Week 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (77):
- United States (18):
  - Tucson, Arizona
  - Artesia, California
  - Jacksonville, Florida
  - Dunwoody, Georgia
  - Idaho Falls, Idaho
  - Aurora, Illinois
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Naperville, Illinois
  - Overland Park, Kansas
  - Livonia, Michigan
  - Chesterfield, Missouri
  - Margate City, New Jersey
  - Trenton, New Jersey
  - Cincinnati, Ohio
  - Bristol, Tennessee
  - San Antonio, Texas
  - Richmond, Virginia
- Czechia (9):
  - Benešov
  - Holice V Cechach
  - Kladno
  - Mladá Boleslav
  - Olomouc
  - Prague
  - Trutnov
  - Ústí nad Orlicí
  - Zlín
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Tampere
  - Turku
- Germany (8):
  - Berlin
  - Bochum
  - Chemnitz
  - Dresden
  - Frankfurt
  - Görlitz
  - Leipzig
  - Nuremberg
- Poland (10):
  - Krakow
  - Leszno
  - Lublin
  - Niemodlin
  - Ostrowiec Świętokrzyski
  - Skierniewice
  - Sroda Wlkp
  - Starachowice
  - Warsaw
  - Zakopane
- Slovakia (7):
  - Banská Bystrica
  - Bojnice
  - Bratislava
  - Lučenec
  - Prešov
  - Šamorín
  - Žilina
- South Africa (6):
  - Bloemfontein
  - Cape Town
  - Durban
  - Lyttleton
  - Pretoria
  - Randburg
- United Kingdom (12):
  - Bath
  - Birmingham
  - Blackpool
  - Blantyre
  - Chippenham
  - Edinburgh
  - Glasgow
  - Harrow
  - Hinckley
  - Newport
  - Nottingham
  - Woolpit

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985